CLINICAL TRIAL: NCT03972917
Title: Long-term Observation of Symptomatic Women With Uterine Fibroids Who Have Been Treated With Ulipristal Acetate: Findings on Symptomatology, Morphological Structure, Endometrial Patterns
Brief Title: Observation of Long-term Effects on Endometrium and Uterine Fibroids in Women With Ulipristal Acetate Therapy
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Prof. Pasquale De Franciscis, Associate Professor, University of Campania Luigi Vanvitelli
Other Study IDs: N.595
Record Dates: First submitted 2019-05-21; First posted 2019-06-04 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Myoma; Uterine Bleeding, Dysfunctional; Uterine Bleeding Heavy; Dysmenorrhea; Endometrium Hyperplasia
Keywords: ulipristal acetate; myoma; leiomyoma; endometrial patterns; symptomatology
MeSH Terms: conditions — Myoma; Metrorrhagia; Dysmenorrhea; Endometrial Hyperplasia; Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ulipristal acetate based therapy: Fertile women under ulipristal acetate treatment
  Interventions: Diagnostic Test: Transvaginal ultrasonographic examination

INTERVENTIONS:
Diagnostic Test: Transvaginal ultrasonographic examination — Evaluation of endometrial thickness; myoma size and volume

SUMMARY:
A prospective observational study on italian women undergoing ulipristal acetate (uPa) therapy for symptomatic myomas and its impact on symptomatology and moreover on myomas architecture. We also evaluate changes in the endometrial pattern of selected women.

ELIGIBILITY:
Inclusion Criteria:

* number of myomas from 1 to 4
* heavy menstrual bleeding
* conservative treatment request

Exclusion Criteria:

* concurrent endometrial pathology
* post-menopausal status
* hepatic pathology
* endocrine or metabolic disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Italian fertile women who are eligible for conservative treatment for uterine fibroids
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Dysmenhorrea (VAS score) | 12 months
Endometrial thickess (mm) | 12 months
Myoma's diameter (mm) | 12 months

SECONDARY OUTCOMES:
Live birth rate (LBR) | 12 months
  Live birth rate if women conceived spontaneously or through ARTs after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Riemma, MD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Department of Woman, Child and General and Specialized Surgery, University of Campania "Luigi Vanvitelli", Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided